CLINICAL TRIAL: NCT06733220
Title: Assessment of Balance in the Strabismic Patient Undergoing Strabismus Surgery
Brief Title: Balance in the Strabismic Patient Undergoing Strabismus Surgery
Acronym: BASS
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Salerni Annabella, Principal investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 7161
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Strabismus
Keywords: Strabismus; Balance; Risk of falling; Quality of life
MeSH Terms: conditions — Strabismus | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- STR-CONG: Patients with congenital strabismus will undergo a comprehensive eye and orthoptic examination and balance test before strabismus surgery at 30 days after surgery, at 90 days after surgery, and at 180 days after surgery.
  Interventions: Procedure: Surgery for strabismus
- STR-ACQ: Patients with acquired strabismus will undergo a comprehensive eye and orthoptic examination and balance test before strabismus surgery, at 30 days after surgery, at 90 days after surgery, and at 180 days after surgery.
  Interventions: Procedure: Surgery for strabismus

INTERVENTIONS:
Procedure: Surgery for strabismus — Patients will undergo surgery to correct strabismus, congenital or acquired

SUMMARY:
Strabismus is a clinical condition characterized by the failure of the visual axes of the two eyes to align on the stared object. There are many possible causes of strabismus, but it can be divided into two main groups: concomitant strabismus, which is characterized by an almost equal angle of deviation in all positions of gaze, and incomitant or paralytic strabismus, which is characterized by a deficit of ocular motility in one or more directions of gaze. Depending on the age of onset, congenital strabismus and acquired strabismus are distinguished. Concomitant strabismus and incomitant strabismus can occur in both plastic age and adults. They are accompanied by diplopia or confusion if they arise in adulthood; there is no diplopia if they arise in plastic age due to cortical compensation mechanisms such as suppression or abnormal retinal matching. Causes of incomitant strabismus in adults can be: decompensation of a preexisting heterophoria; acute incomitant strabismus; injury to fusional centers. Paralytic incomitant strabismus is characterized by a reduction in the force developed by one or more muscles of an eye. Among incomitant strabismus, restrictive strabismus represent clinical pictures of very different etiology united by a single distinguishing feature: the existence of a mechanical obstacle to the free movement of the bulb in the orbit that prevents or reduces the excursion of the eye in one or more directions of gaze.

In about 4% of the young population, the sensory and/or motor pathways are not adequately developed, resulting in misalignment of the visual axes and strabismus. Eye surgery for strabismus is one of the most widely used treatment methods.

Only a few studies in the literature have analyzed changes in postural control after strabismus surgery and on a limited number of patients.

A French study evaluated the effect of surgery on postural control in children with strabismus, concluding that eye surgery affects the somatosensory properties of extraocular muscles, leading to improved postural control and that binocular visual perception could affect the whole body.

DETAILED DESCRIPTION:
Patients belonging to the UOC Ophthalmology, the UOS Diagnosis and Treatment of Ocular Motility Disorders and the Pediatric Ophthalmology Outpatient Clinic, Fondazione Policlinico Universitario A. Gemelli IRCCS in Rome who meet the inclusion criteria will be recruited. Patients will be divided into two groups according to the nature of strabismus (congenital or acquired). All patients, regardless of the nature of strabismus, will undergo a complete ophthalmologic and orthoptic examination and balance examination before strabismus surgery (baseline, T0), at 30 days after surgery (T1), at 90 days after surgery (T2), and at 180 days after surgery (T3).

All patients will undergo clinical evaluation and assessment of balance and fall risk at all assessment timepoints

ELIGIBILITY:
Inclusion Criteria:

* Age between 16 and 65 years;
* Presence of congenital strabismus or acquired strabismus in the care of the Ophthalmology OU, the Diagnosis and Treatment of Ocular Motility Disorders OU, and the Pediatric Ophthalmology Outpatient Clinic
* Ability to maintain balance safely for at least 180 seconds;
* In case of adult patient, Ability to understand and sign informed consent
* In case of minor patient, Ability to understand and sign the assent for participation in the study and consent from the parent

Exclusion Criteria:

* Presence of diplopia associated with nystagmus;
* Presence of psychomotor and cognitive delay, as assessed by the Mini Mental State Examination (adjusted score < 24);
* Noncooperation of the patient;
* Inability to provide informed consent, in the case of adult patients.
* Inability to provide consent in case of minor patients, or consent from parents.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with strebismus, congenital or acquired, who will have surgery for surgical correction of strabismus during the study period will be included.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Dynamic balance | Change from Baseline Dynamic Balance at 30, 90 and 180 days
  Dynamic balance will be assessed using a robotic platform. Specifically, the reduction in the displacement of the center of pressure under dynamic conditions will be evaluated

SECONDARY OUTCOMES:
Cover/Uncover test | Change from Baseline Cover/Uncover test at 30, 90 and 180 days
  It is a useful test to assess some characteristics of strabismus. It is always performed for both distance (6 m) and near (33 cm). The cover/uncover test is performed by occluding one of the two eyes with a screen for a few seconds and then uncovering it again allowing binocular vision, then performing the same maneuver on the other eye. Next, the alternating cover test is performed, which consists of covering first one eye and then the other with a screen, without allowing both eyes to see at the same time.
Cover test with prisms | Change from Baseline Cover test with prisms at 30, 90 and 180 days
  The test allows measurement of the angle of strabismus and is performed by sliding a slat of Berens prisms in front of either eye. The cover-test is repeated by sliding the prism bar and observing the amount of movement the deviated eye makes to take fixation. They will decrease, increasing the power of the prism, until they are cancelled. The prism that cancels the movement corresponds to the magnitude, in prism diopters, of the deviation angle.
Irvine test | Change from Baseline Irvine test at 30, 90 and 180 days
  The test consists of placing an externally based prism of 4 prism diopters in front of one eye. If there is convergence movement due to the disparity of image presentation to the two eyes, there is fusion movement, and if such movements are present for near (33 cm) and far (6 m and beyond), there is normal binocular vision. Otherwise, fusional motion will be absent.
Angle measurement in the various positions of gaze | Change from Baseline angle measurement at 30, 90 and 180 days
  The method generally employed for this measurement is the screen test (cover test) in conjunction with a vertical or horizontal prism bar. Ocular deviation should be assessed in the following positions of gaze:
  * primary position, with head erect and looking straight ahead;
  * 4 secondary positions, are straight down, straight up, horizontally right and left;
  * 4 tertiary positions, are the oblique positions (up right and left, down right and left) Evaluation of these nine positions of gaze, referred to as diagnostic positions, provides a complete picture of alterations in the function of various muscles.
Bagolini's Streaked Glasses | Change from Baseline Bagolini's Streaked Glasses at 30, 90 and 180 days
  Streaked glasses are flat lenses with thin streaks along a meridian. On each glass is a mark called the striated glass axis, which indicates the orientation of the light streak seen by the patient. The test is performed for near (33 cm) and far (6 m). It can identify:
  a normal retinal match if there is no bulb deviation or an abnormal retinal match if tropic motion is detected in the cover-uncover test.
  Complete suppression of the deviated eye. This is a condition prevalent in wide-angle strabismus.
  suppression scotoma.
  - diplopia disparity of fixation.
Worth lights | Change from Baseline Worth lights at 30, 90 and 180 days
  This test consists of four lights, 2 green, 1 red and 1 white. It can be performed for both distance and near; the patient being tested must stare at the four lights while wearing a pair of anaglyphic glasses (red-green lenses). Since the lights are complementary to the filters placed in front of the patient's eyes, he will see red light through the red filter and green light through the green filter. The patient can see:
  * four lights (one red, two green and a fourth red or green depending on ocular dominance), indicating normal retinal matching or abnormal retinal matching;
  * three green lights or two red lights in case of suppression;
  * five lights (two red and three green) in case of diplopia.
Lang's test | Change from Baseline Lang's test at 30, 90 and 180 days
  Lang's test consists of the presentation of a card in which there are random stimuli printed with a panographic system, that is, with small cylinders oriented so that each is perceived by only one eye. The disparities proposed in Lang's first test range from 600 to 1200 arc seconds, specifically the star and the car have a disparity of 600 arc seconds, while the cat has a disparity of 1200 arc seconds.
TNO test | Change from Baseline TNO test at 30, 90 and 180 days
  TNO test This test splits images with a red and green complementary color glasses. The parts of the images displayed stimulate the eyes separately: the red parts of the images are seen only by the eye with the red glass; the green parts only by the eye with the green glass. In binocular combination, parts of these images stimulate different retinal areas and are seen in relief. This test provides images with gradations of up to 15 arc seconds.
Red Glass test | Change from Baseline Red Glass test at 30, 90 and 180 days
  A red glass is placed in front of one of the eyes and a bright vision is presented to the patient, which is arranged in the various positions of gaze. If there is a deficit, the patient sees two lights, one white and one red, indicative of diplopia. The test is based on finding the direction of gaze in which diplopia is greatest. First, it must be ascertained whether diplopia is also present in primary gaze; then it is assessed whether it is greater in the right or left version and finally whether it is such, or increases, in upward or downward gaze. Another important finding is whether diplopia is horizontal and/or vertical. Once the direction of gaze in which the two fixation view images are furthest apart is established, the diagnosis will have been limited to only two muscles (one in each eye). Keeping in mind that the image of the eye with the muscle deficit is always the one farthest from the patient, it will be easy to arrive at an exact determination of the deficit muscle.
Prism Adaptation Test (PAT) | Change from Baseline PAT at 30, 90 and 180 days
  The PAT aims to assess whether the phenomenon of prism compensation (abnormal fusion movements) occurs. Prisms that best neutralize the deviation are placed in front of the eyeglass; after a longer or shorter observation period, three possibilities may occur:
  1. the angle does not change, the patient does not compensate for the prisms;
  2. As the angle of deviation increases, the patient compensates for the prisms; we are probably in the presence of abnormal fusion movements. These may be: poorly rooted, very rooted, apparent;
  3. the angle of deviation decreases (rare occurrence).
Prism Progressive Test (PPT) | Change from Baseline PPT at 30, 90 and 180 days
  The PPT is used to evaluate, in cases of prism compensation, the radication of MFAs. Prisms of magnitude greater than the deflection angle are placed in front of them and it is observed whether they are compensated or not.
Binocular field of gaze for diplopia | Change from Baseline Binocular field of gaze for diplopia at 30, 90 and 180 days
  This examination involves evaluating areas of diplopia and single vision within the visual field. It is useful for tracking the progress of paralysis or the effect of surgery. It is performed with Goldmann's perimeter in binocular vision. It is done by placing the subject seated in front of the perimeter, a light sight is presented that moves over the various meridians, the patient is asked to follow it with his or her eyes, and an assessment is made of where the subject sees double the light projected by the perimeter and where there may be areas of single vision. Areas of diplopia and single binocular vision are mapped in the appropriate perimetry diagrams.
Silver Index (SI) | Change from Baseline SI at 30, 90 and 180 days
  The SI is an objective test conducted through a robotic platform that can identify the risk of falling. It consists of seven domains: (i) static balance, (ii) dynamic balance, (iii) reactive balance, (iv) sensory integration, (v) stability limits, (vi) sit-to-stand, and (vii) gait speed.
  The platform returns a fall risk ranging from 0% to 100%: higher values indicate higher fall risk

CONTACTS AND LOCATIONS:
Overall Officials: Annabella Salerni, MD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No